CLINICAL TRIAL: NCT03383445
Title: Transcatheter Aortic Valve Replacement Versu Surgical Aortix Valve Replacement for Treating Elderly Patients With Severe Aortic Stenosis and Small Aortic Annuli: A Prospective Randomized Study The VIVA Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec (Other)
Responsible Party: Principal Investigator, Josep Rodes-Cabau, MD, Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec
Organization: Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VIVA
Record Dates: First submitted 2017-06-28; First posted 2017-12-26 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Degenerative Aortic Valve Disease; Aortic Stenosis; Aortic Regurgitation
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Insufficiency

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in a 1:1 fashion to either TAVR or SAVR
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TAVR (Other): The TAVR procedure will be performed following the standards of each participating center. No restriction or specific recommendation will be given regarding the approach, general vs. local abesthesia, Imaging guidance during the TAVR procedure, and post-procedural TAVR management.
  Interventions: Procedure: Edwards; Procedure: CoreValve; Procedure: Acurate neo
- SAVR (Other): SAVR procedure will be performed using standard techniques, with no limitation in terms of type and size of the valve prosthesis or surgical procedure (e.g. enlargement of the aortic root).
  Interventions: Procedure: Standard

INTERVENTIONS:
Procedure: Edwards — The TAVR procedure will be performed with the Edwards SAPIEN XT or SAPIEN 3 valve (20, 23 or 26 mm).
  Arms: TAVR
Procedure: CoreValve — The TAVR procedure will be performed with the CoreValve Evolut R valve system (23 or 26 mm).
  Arms: TAVR
Procedure: Acurate neo — The TAVR procedure will be performed with the ACURATE neo aortic valve.
  Arms: TAVR
Procedure: Standard — The choice of the type and size of valve, utilization of additional procedures such as root enlargement will be left at the discretion of heart team of the treating the patient.
  Arms: SAVR

SUMMARY:
To date, no formal, randomized, prospective, head-to-head comparisons of surgical aortic valve replacement (SAVR) versus transcatheter aortic valve replacement (TAVR) have been undertaken in the severe aortic stenosis (AS) population with small aortic annuli. Objectives of the present study are to compare the hemodynamic performance (incidence of severe PPM and ≥ moderate AR) and clinical outcomes (death, stroke, major or life threatening bleeding) between TAVR and SAVR in patients with severe AS and small aortic annuli.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized open-label trial including patients with severe AS and small aortic annulus (mean aortic annuli diameter ˂23mm and minimal diameter ≤21.5mm, evaluated by 3D-CT or 3D-TEE). Patients will be randomized in a 1:1 fashion to either TAVR or SAVR. The TAVR procedure will be performed with the ACURATE neo Aortic Valve, the Edwards SAPIEN 3 valve (20, 23 or 26mm) or the CoreValve Evolut R or Evolut PRO valve system (23 or 26 mm).New iterations of these valve models may also be included. The SAVR procedure will be performed using standard techniques, with no limitation in terms of type and size of the valve prosthesis or surgical procedure (e.g. enlargement of the aortic root). For both TAVR and SAVR, the choice of the type and size of valve, access route (for TAVR), utilization of additional procedures such as root enlargement will be left at the discretion of heart team of the site treating the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥65 years-old diagnosed with severe AS (defined as: jet velocity ≥ 4.0 m/s or mean gradient ≥ 40 mmHg or velocity ratio <0.25 AND aortic valve area ≤ 1.0 cm2 or aortic valve area index ≤ 0.6 cm2/m2; OR mean gradient >30 mmHg AND aortic valve area ≤ 1.0 cm2 or aortic valve area index ≤ 0.6 cm2/m2 AND >1200 Agatston units for women or >2000 Agatston units for men as determined by non-contrast CT).
* Small aortic annulus defined as a mean aortic annulus diameters ˂23 mm and a minimal aortic annulus diameter of ≤21.5 mm as measured by 3D-computed tomography (CT) and/or 3D-transesophageal echocardiography (TEE).

Exclusion Criteria:

* Prohibitive surgical risk as determined by the Heart Team
* Porcelain aorta
* Aortic root dilatation >45 mm
* Coronary artery disease (CAD) not treatable by percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG), or SYNTAX score >32 (in the absence of prior revascularization) or severe left main disease
* Non-calcific aortic stenosis
* Severe mitral regurgitation
* Moderate-to-severe tricuspid regurgitation requiring surgical repair
* Prior surgical valve in aortic position

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-08-08 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Valve performance: rate of prothesis-patient mismatch (PPM) and/or aortic regurgitation (AR) | 60 days
  Severe PPM [defined as an indexed aortic valve area ≤0.65 cm2/m2 ] and/or ≥moderate AR [Valve Academic Research Consortium-2 (VARC-2) definition].

SECONDARY OUTCOMES:
Rate of PPM | 60 days, 1 year and 5 years
  Rate of moderate or severe PPM
Rate of AR | 60 days, 1 year and 5 years
  Rate of moderate or severe AR
Combined endpoints: rate of AR or PPM | 1 year and 5 years
  Moderate or severe AR or severe PPM
Transvalvular gradient | 60 days, 1 year and 5 years
  Mean transvalvular gradient
Combined endpoints: LVEF and LV | 60 days, 1 year and 5 years
  Changes in LVEF and LV hypertrophy
Mortality | 30 days, 1 year and 5 years
  Death
Stroke | 30 days, 1 year and 5 years
  Stroke (Valve Academic Research Consortium-2 (VARC-2) definition)
Bleeding | 30 days, 1 year and 5 years
  Major or life threatening bleeding
Rate of new atrial fibrillation | 30 days, 1 year and 5 years
  Rate of new-onset atrial fibrillation
Combined Safety endpoint | 30 days, 1 year and 5 years
  Death, stroke, major/life threatening bleeding
Cardiac re-hospitalization | 30 days, 1 year and 5 years
  Need for cardiac re-hospitalization
Day of hospital stay | For the duration of hospital stay
  Length of the hospitalization for the TAVR or SAVR procedure
Quality of life | 30 days, 60 days, 1 year and 5 years
  Questionnaire, visual scale
Exercise capacity | 60 days, 1 year and 5 years
  Exercise capacity as evaluated by the six-minute walk test

CONTACTS AND LOCATIONS:
Locations (1):
- IUCPQ, Québec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rodes-Cabau J, Ribeiro HB, Mohammadi S, Serra V, Al-Atassi T, Iniguez A, Vilalta V, Nombela-Franco L, Saez de Ibarra Sanchez JI, Auffret V, Forcillo J, Conradi L, Urena M, Moris C, Munoz-Garcia A, Paradis JM, Dumont E, Kalavrouziotis D, Maria Pomerantzeff P, Rosa VEE, Pezzute Lopes M, Sureda C, Diaz VAJ, Giuliani C, Avvedimento M, Pelletier-Beaumont E, Pibarot P; VIVA (Transcatheter Aortic Valve Replacement Versus Surgical Aortic Valve Replacement for Treating Elderly Patients With Severe Aortic Stenosis and Small Aortic Annuli) Trial Investigators. Transcatheter or Surgical Aortic Valve Replacement in Patients With Severe Aortic Stenosis and Small Aortic Annulus: A Randomized Clinical Trial. Circulation. 2024 Feb 27;149(9):644-655. doi: 10.1161/CIRCULATIONAHA.123.067326. Epub 2023 Oct 26. PMID 37883682